CLINICAL TRIAL: NCT04029909
Title: A Phase I Clinical Study of Gimatecan (ST 1481) in Patients With Platinum-resistant or Sensitive Relapsing/Refractory Advanced Ovarian Epithelial Cancer, Fallopian Tube Cancer or Primary Peritoneal Cancer
Brief Title: A Clinical Study of Gimatecan in Advanced Ovarian Epithelial Cancer, Fallopian Tube Cancer or Primary Peritoneal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NTL-LEES-2018-01
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Ovarian Epithelial Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — ST 1481

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gimatecan 0.6mg/m2/d (Experimental): Three or six patients will be treated with the dose of 0.6mg/m2/d for once a day for 5 consecutive days of Gimatecan. DLT will be observed within 28 days after administration.
  Interventions: Drug: Gimatecan 0.6mg/m2/d
- Gimatecan 0.8mg/m2/d (Experimental): Three or six patients will be treated with the dose of 0.8mg/m2/d for once a day for 5 consecutive days of Gimatecan. DLT will be observed within 28 days after administration.
  Interventions: Drug: 0.8mg/m2/d
- Gimatecan 0.4mg/m2/d (Experimental): Three or six patients will be treated with the dose of 0.4mg/m2/d for once a day for 5 consecutive days of Gimatecan. DLT will be observed within 28 days after administration.
  Interventions: Drug: 0.4mg/m2/d

INTERVENTIONS:
Drug: Gimatecan 0.6mg/m2/d — 0.6mg/m2/d for once a day for 5 consecutive days of Gimatecan
  Arms: Gimatecan 0.6mg/m2/d
Drug: 0.8mg/m2/d — 0.8mg/m2/d for once a day for 5 consecutive days of Gimatecan
  Arms: Gimatecan 0.8mg/m2/d
Drug: 0.4mg/m2/d — 0.4mg/m2/d for once a day for 5 consecutive days of Gimatecan
  Arms: Gimatecan 0.4mg/m2/d

SUMMARY:
This is a Phase 1, open-label, dose-escalation ,and multidose study, aiming to investigate the safety, tolerability and pharmacokinetics of Gimatecan in Advanced Ovarian Epithelial Cancer, Fallopian Tube Cancer or Primary Peritoneal Cancer. To explore the dose-limiting toxicity (DLT) and the maximum tolerable dose (MTD) of oral administration of Gimatecan capsules 5 consecutive days, every 28 days.

DETAILED DESCRIPTION:
The clinical trial is used the traditional 3 +3 design and conducted in two dose groups, 0.6mg/m2/d and 0.8mg/m2/d, with an improved dose escalation design. The initial dose is 0.6mg/m2, once a day for 5 consecutive days, every 28 days for a course of treatment. Subjects are assigned to the corresponding dose group according to the order of enrolling. DLT is observed within 28 days of the first dose of Gimatecan. In the absence of DLT as prescribed by the protocol, the next dose group is started until the maximum tolerated dose (MTD) is observed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have stage III or IV ovarian epithelial cancer, fallopian tube cancer or primary peritoneal cancer.
2. Definite histopathological diagnosis.
3. Failed with treatment for taxane/doxorubicin and platinum.
4. Must have measurable disease with at least 1 unidimensional measurable lesion base on RECIST1.1. When evaluating the efficacy of patients with CA125 level, CA125 abnormalities caused by other reasons should be excluded. According to the Gynecologic Cancer Intergroup-GCIG standard, the baseline serum CA125 level of patients within 2 weeks before treatment should be ≥2 upper limit of normal.
5. Age between 18-65(inclusive).
6. ECOG（Eastern Cooperative Oncology Group） performance status of 0 or 1.
7. To estimated life expectancy of at least 3 months.
8. Appropriate blood routine, liver and kidney function.
9. No allergic history of camptothecin.
10. Patients who are able to take strict contraceptive measures during the trial and within 4 months after the end of the trial.
11. The patients are able to swallow and maintain oral medication.
12. More than 4 weeks from the end of previous surgery, chemotherapy, radiotherapy (non-pelvic and peritoneal sites) and targeted therapy before the study and the body had recovered (the treatment-related toxicity grade is no more than grade 1, except for hair loss and pigmentation).
13. Patients voluntarily give written informed consent to participate in the study.

Exclusion Criteria:

1. The patients are treated with irinotecan or topotecan or with any topoisomerase I inhibitor regimen prior to enrollment.
2. Patients who use other experimental drugs or conducted other clinical trials at the same time within 30 days before participate in the study.
3. To received radiotherapy of pelvic cavity and abdomen.
4. Smoking more than 5 cigarettes per day in the past year.
5. Suspected or real alcohol dependence with an average alcohol intake of more than 2 units per day for 3 months.
6. Active infection.
7. patients with the history of gastrointestinal surgery or that may change drug absorption and activity in the body.
8. Serious cardiovascular disease, including Ⅱ magnitude abnormal cardiac function.
9. having a clear history of neuropathy or mental disorders (including epilepsy or dementia).
10. Human immunodeficiency virus(HIV) positive, untreated active hepatitis.
11. Suffering from other malignant tumors other than this diseases in 5 years, except for basal cell carcinoma of skin, skin squamous cell carcinoma, primary cervical carcinoma and breast cancer without recurrence and metastasis after radical operation.
12. Brain metastasis.
13. Female with pregnant or lactating.
14. Patients who are considered unsuitable to participate in the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 12 (Estimated)
Dates: Start 2019-07-11 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity(DLT) | 28 days after first dose
  Adverse events of level 3 or above related to the study drug occurring within 28 days after the first dose as assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
Maximal tolerable dose(MTD) | 28 days after first dose
  DLT occurs in less than 1/6 subjects, this lower dose is defined as MTD.

OTHER OUTCOMES:
The overall response rate(ORR) | through study completion, an average of 2 years
  The proportion of subjects who achieve the optimal objective response rate(PR or CR).
AUC(0-t) | 28 days after first dose
  Area under curve 0-t
Cmax | 28 days after first dose
  Peak concentration
Tmax | 28 days after first dose
  Peak concentration
T1/2 | 28 days after first dose
  Half life

CONTACTS AND LOCATIONS:
Overall Officials: Hong Zheng, MD, Study Director — Beijing Tumor Hospital
Locations (1):
- Beijing Tumor Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No